CLINICAL TRIAL: NCT05907447
Title: A Retrospective Study on Extranodal Lymphoma or Lymphoma of Rare Pathological Types
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Fujian Medical University Union Hospital (Other); Peking University Third Hospital (Other); Peking University People's Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); The Second Affiliated Hospital of Dalian Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Henan Provincial People's Hospital (Other); Hunan Cancer Hospital (Other); Henan Cancer Hospital (Other Government); The First Hospital of Jilin University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Affiliated Hospital of Nantong University (Other); The First Affiliated Hospital of Xiamen University (Other); Shandong Provincial Hospital (Other Government); Shanxi Province Cancer Hospital (Other); RenJi Hospital (Other); Beijing Friendship Hospital (Other); West China Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Tongji Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sun Yat-sen University (Other); Chongqing University Cancer Hospital (Other); Anhui Provincial Cancer Hospital (Other); The General Hospital of Northern Theater Command (Other); Qilu Hospital of Shandong University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Wuhan TongJi Hospital (Other); General Hospital of Ningxia Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Anshan Central Hospital (Other); Hainan Cancer Hospital (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Other Study IDs: EXPECT-01
Record Dates: First submitted 2023-05-01; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma; Extranodal Lymphoma; Diffuse Large B Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Marginal Zone Lymphoma; Mucosa-Associated Lymphoid Tissue Lymphoma; NK/T-Cell Lymphoma, Nasal and Nasal-Type; Intravascular Large B-Cell Lymphoma
Keywords: LYMPHOMA; EXTRANODAL
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions need to be specified for this study — No interventions need to be specified for this study

SUMMARY:
The aim of this study is to retrospectively collect clinical information on patients with extranodal or rare lymphomas, and to explore the best treatment strategy for these lymphomas in the real-world population.

DETAILED DESCRIPTION:
Lymphoma is a highly common malignant tumor in Asia. For specific extra-abdominal sites or rare pathological subtypes of lymphoma, traditional chemotherapy protocols often cannot provide satisfactory results for patients. This study aims to retrospectively collect clinical information on patients with extranodal lymphoma or rare pathological subtype lymphoma, including the distribution of involved sites, clinical and molecular characteristics of different lymphoma subtypes, clinical treatment protocols, and prognosis, to explore the best treatment strategy for these lymphomas in the real-world population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (including 18 years old).
2. Patients newly diagnosed with non-Hodgkin lymphoma with extranodal involvement, whether it is primary, secondary, or cannot be determined; Or patients newly diagnosed with non-Hodgkin lymphoma of rare pathological types, including IVLBCL, SMZL, ALCL, AITL, MALTL.
3. Patients who have received systematic clinical treatment.
4. Patients with measurable lesions, at least containing one effective evaluation of efficacy.

Exclusion Criteria:

1. Patients who only receive supportive treatment.
2. Patients who cannot obtain effective evaluation data of efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically confirmed diagnosis of non-Hodgkin lymphoma with extranodal involvement or non-Hodgkin lymphoma of rare pathological types attending participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline up to data cut-off (up to approximately 1 year)
  Overall Survival (OS) will be defined from the start date of therapy to the date of death from any cause.
Progression Free Survival (PFS) | Baseline up to data cut-off (up to approximately 1 year)
  Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.

SECONDARY OUTCOMES:
Clinical characteristics form | Baseline up to data cut-off (up to approximately 1 year)
  Clinical characteristics from data filled into registry forms by physicians and data managers, including but not limited to values of lactate dehydrogenase, clinical stage, performance status, age ≥ 60 years and number and location of extranodal localizations.
Biological characteristics form | Baseline up to data cut-off (up to approximately 1 year)
  Biological characteristics from data filled into registry forms by physicians and data managers, such as immunohistochemical differences and genetic mutation characteristics of non-hodgkin´s lymphomas.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided